CLINICAL TRIAL: NCT06746441
Title: Effect of Psilocybin Only and Psilocybin Assisted Cognitive Behavioral Therapy in the Management of Major Depressive Disorder and Associated Metabolic, Immune, Inflammatory, Neuroplasticity and Electrical Activity Markers: a Randomized Controlled Trial
Brief Title: Effect of Psilocybin Only and Psilocybin Assisted Cognitive Behavioral Therapy in the Management of Major Depressive Disorder and Associated Metabolic, Immune, Inflammatory, Neuroplasticity and Electrical Activity Markers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/011
Record Dates: First submitted 2024-12-09; First posted 2024-12-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder
Keywords: Psilocybin; Cognitive Behavioral Therapy (CBT); Randomized Controlled Trial; Psychedelic Therapy; Inflammatory Markers
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psilocybin; psilocin; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment (The study has four distinct intervention groups: Control, Psilocybin Therapy, CBT, and Psilocybin-assisted CBT.)
Who Masked: Participant
Masking Description: Randomized (Random allocation will be performed using a simple lottery method.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Psilocybin Therapy Group (Experimental): Participants will receive two oral doses of psilocybin (5-6 grams per dose), administered six weeks apart. Each session will occur in a controlled environment with medical monitoring until the hallucination phase subsides. Participants will continue their routine antidepressant medications during the study.
  Interventions: Drug: Psilocybin
- Control Group (No Intervention): Participants will continue their routine antidepressant medications (e.g., SSRIs such as citalopram, escitalopram, or sertraline) without any additional intervention.
- Cognitive Behavioral Therapy (CBT) Group (Active Comparator): Participants will undergo 8-10 structured sessions of Cognitive Behavioral Therapy over six weeks. Each session will last approximately 90 minutes, focusing on restructuring negative thought patterns and addressing depression symptoms. Participants will continue their routine antidepressant medications during the study.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Psilocybin-Assisted CBT Group (Active Comparator): Participants will receive both psilocybin therapy and Cognitive Behavioral Therapy. Psilocybin will be administered in two oral doses (5-6 grams per dose), six weeks apart, with medical monitoring during sessions. In addition, participants will undergo 8-10 CBT sessions over six weeks. Routine antidepressant medications will be continued.
  Interventions: Drug: Psilocybin; Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: Psilocybin — Psilocybin is a naturally occurring serotonergic psychedelic compound found in Psilocybe mushrooms. It is metabolized in the body into its active form, psilocin, which has a high affinity for serotonin 5-HT2A receptors. This enables psilocin to bypass the default serotonin pathway, producing antidepressant effects.
  For this study:
  Psilocybin will be administered orally in a dose of 5-6 grams per session. Each participant in the Psilocybin and Psilocybin-assisted CBT arms will receive two sessions spaced six weeks apart.
  The therapy will be conducted in a controlled hospital setting with medical monitoring during the session to ensure safety until the hallucination phase subsides.
  Psilocybin will be added to routine antidepressant medication.
  Other Names: Psilocin (the active form of psilocybin metabolized in the body)
  Arms: Psilocybin Therapy Group; Psilocybin-Assisted CBT Group
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive Behavioral Therapy (CBT) is a structured, time-limited psychotherapy aimed at alleviating symptoms of depression. It involves addressing negative thoughts and behavioral patterns through the following steps:
  Identifying troubling life situations. Recognizing thoughts, emotions, and beliefs about those situations. Identifying negative or inaccurate thinking patterns. Restructuring those thoughts into positive and realistic perspectives.
  In this study:
  CBT will consist of 8-10 structured sessions, each lasting approximately 90 minutes.
  Participants will attend therapy sessions twice weekly over a six-week period. The intervention will be delivered by trained psychotherapists in a controlled hospital setting.
  Routine antidepressant medications will be continued alongside CBT.
  Arms: Cognitive Behavioral Therapy (CBT) Group; Psilocybin-Assisted CBT Group

SUMMARY:
This randomized controlled clinical trial evaluates the effectiveness of psilocybin and psilocybin-assisted cognitive behavioral therapy (CBT) in the management of Major Depressive Disorder (MDD). The study aims to compare the effects of psilocybin-only therapy, CBT, and psilocybin-assisted CBT on depression symptoms, neurochemical markers, inflammatory markers, and neuroplasticity in individuals with MDD. Participants will continue their routine depression medications and will be assessed for changes in depression scores, biochemical markers, and brain activity patterns using validated tools and tests.

DETAILED DESCRIPTION:
This single-masked randomized controlled trial investigates novel therapeutic interventions for Major Depressive Disorder (MDD). MDD is a leading cause of disability worldwide, with a significant proportion of patients being treatment-resistant or showing only partial response to conventional antidepressants. Emerging evidence suggests that psilocybin, a serotonergic psychedelic, has potential as a rapid-acting antidepressant.

The study will recruit 60 participants meeting DSM-V criteria for MDD, randomized into four groups:

Control group (Conventional therapy only), Psilocybin therapy group, Cognitive Behavioral Therapy (CBT) group, and Psilocybin-assisted CBT group. Participants will receive interventions over 10 weeks, with psilocybin administered in two heroic doses six weeks apart, and CBT delivered in 8-10 structured sessions. Biochemical and neurochemical markers such as CD4/CD8 ratio, TNF-α, IL-6, BDNF, and oxytocin will be measured, along with inflammatory markers (resistin and visfatin). Depression scores will be assessed using scales like HAM-D, MADRS, and BDI. EEG recordings will evaluate changes in brain activity pre- and post-intervention.

The primary objective is to assess improvements in depression symptoms, while secondary objectives include evaluating changes in immune, inflammatory, and neurochemical markers and EEG activity. Data will be analyzed using ANOVA with Tukey's post-hoc tests to determine statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-70 years.
* Diagnosed with Major Depressive Disorder (MDD) according to DSM-V criteria.
* Active depressive symptoms as indicated by a score > 16 on the Hamilton Depression
* Rating Scale (HAM-D) over the preceding two weeks.
* Female participants of childbearing potential must be using a highly effective form of contraception and willing to maintain contraceptive use throughout the study period.
* Participants must have been taking one SSRI antidepressant (e.g., citalopram, escitalopram, fluoxetine) for at least 6 weeks with at least 75% adherence.

Exclusion Criteria:

* Resting blood pressure >140/90 (average of four separate measurements).
* Risk of suicidal tendencies as indicated by a score of 3 or higher on item 3 of the HAM-D scale.
* Use of multiple SSRIs or any antidepressant not specified in the inclusion criteria.
* Presence of concurrent psychiatric disorders (e.g., bipolar disorder, schizophrenia).
* Use of psychedelics or ketamine within the last 12 months.
* Pregnancy, breastfeeding, or attempting to conceive.
* History of substance abuse or alcohol use in the last 6 months.
* Cardiovascular conditions (e.g., hypertension, stroke history).
* History of seizures or epilepsy.
* Diabetes (especially insulin-dependent).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Depression Scores (Hamilton Depression Rating) | Baseline, Week 6 (end of the first psilocybin session), and Week 10 (end of intervention).
  Assessment of changes in depression scores using the Hamilton Depression Rating Scale (HAM-D), a clinician-administered tool for evaluating the severity of depression.
  Unit of Measure: Points on the HAM-D scale. The HAM-D consists of 17 items, each assessing a specific depressive symptom. Each item is rated on a 0-4 or 0-2 scale, depending on the item. The total score ranges from 0 to 52. Higher scores indicate greater severity of depressive symptoms.
  0-7: Normal 8-13: Mild depression 14-18: Moderate depression 19-22: Severe depression
  * 23: Very severe depression
Change in Depression Scores (Montgomery-Åsberg Depression Rating Scale) | Baseline, Week 6 (end of the first psilocybin session), and Week 10 (end of intervention).
  Assessment of changes in depression scores using the Montgomery-Åsberg Depression Rating Scale (MADRS), a clinician-administered scale for evaluating depressive symptom severity.
  Unit of Measure: Points on the MADRS scale.
  The MADRS consists of 10 items, each assessing a specific depressive symptom. Each item is rated on a 0-6 scale. The total score ranges from 0 to 60. Higher scores indicate greater severity of depressive symptoms.
  0-12: Normal 13-19: Mild depression 20-34: Moderate depression
  * 35: Severe depression
Change in Depression Scores (Beck Depression Inventory) | Baseline, Week 6 (end of the first psilocybin session), and Week 10 (end of intervention).
  Assessment of changes in depression scores using the Beck Depression Inventory (BDI), a self-reported measure designed to evaluate the severity of depression symptoms.
  Unit of Measure: Points on the BDI scale.
  The BDI consists of 21 items, each assessing a specific depressive symptom. Each item is rated on a 4-point scale. The total score ranges from 0 to 63. Higher scores indicate greater severity of depressive symptoms.
  0-13: Normal 14-19: Mild depression 20-28: Moderate depression 29-63: Severe depression
Change in Anxiety Scores (Beck Anxiety Inventory) | Baseline, Week 6 (end of the first psilocybin session), and Week 10 (end of intervention).
  Assessment of changes in anxiety scores using the Beck Anxiety Inventory (BAI), a self-reported questionnaire for evaluating the severity of anxiety symptoms.
  Unit of Measure: Points on the BAI scale.
  The BAI consists of 21 items, each assessing a specific anxiety symptom. Each item is rated on a 0-3 scale. The total score ranges from 0 to 63. Higher scores indicate greater severity of anxiety symptoms.
  0-7: Normal 8-15: Mild anxiety 16-25: Moderate anxiety 26-63: Severe anxiety

SECONDARY OUTCOMES:
Change in Brain-Derived Neurotrophic Factor (BDNF) Levels | Baseline, Week 6, and Week 10
  Assessment of changes in serum BDNF levels from baseline to the end of the intervention.
  Unit of Measure: ng/mL.
Change in Oxytocin Levels | Baseline, Week 6, and Week 10
  Assessment of changes in serum oxytocin levels from baseline to the end of the intervention.
  Unit of Measure: pg/mL.
Change in Inflammatory Markers | Baseline, Week 6, and Week 10.
  Evaluation of changes in serum levels of TNF-α, IL-6, resistin, and visfatin to monitor systemic inflammation.
  Unit of Measure: pg/mL or ng/mL, depending on the specific biomarker.
Deviation from Balanced Time Perspective (DBTP) | Baseline, Week 6, and Week 10.
  Measurement of deviation from a balanced time perspective using the Zimbardo Time Perspective Inventory (ZTPI).
  Unit of Measure: ZTPI score.
EEG Pattern Changes | Baseline, Week 6, and Week 10.
  Analysis of changes in EEG activity patterns before and after the intervention, focusing on frequency bands (e.g., Alpha, Beta, Theta, and Delta waves) and their relative power across these bandwidths.
  Unit of Measure: Relative power (percentage or dB).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mahvash Khan, Principal Investigator — Hayat Abad Medical Complex, Peshawar
Locations (1):
- Lady Reading Hospital, Pakistan, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The study will make individual participant data (IPD) available to other researchers after the conclusion of the study. The IPD shared will include anonymized data related to the primary and secondary outcome measures, including depression scores, biochemical markers (e.g., TNF-α, IL-6, BDNF), EEG data, and other relevant clinical and demographic data collected during the trial. The data will be de-identified to ensure participant confidentiality. The data will be shared through an approved data repository or by direct request to the study's primary investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will become available one year after the completion of data analysis (anticipated November 2025). Data will remain accessible for a period of 5 years or until the data usage restrictions are lifted by ethical review.
Access Criteria: The data will be accessible to qualified researchers who meet the following criteria:
  * Ethical approval for data usage from their institution.
  * A research proposal that justifies the use of the data and outlines the planned analysis.
  * Institutional support for data management and ethics review.

REFERENCES:
- [Background] Lee YJ, Lee GW, Seo WS, Koo BH, Kim HG, Cheon EJ. Neurofeedback Treatment on Depressive Symptoms and Functional Recovery in Treatment-Resistant Patients with Major Depressive Disorder: an Open-Label Pilot Study. J Korean Med Sci. 2019 Nov 4;34(42):e287. doi: 10.3346/jkms.2019.34.e287. PMID 31674161
- [Background] MacCallum CA, Lo LA, Pistawka CA, Deol JK. Therapeutic use of psilocybin: Practical considerations for dosing and administration. Front Psychiatry. 2022 Dec 1;13:1040217. doi: 10.3389/fpsyt.2022.1040217. eCollection 2022. PMID 36532184
- [Background] Dodd S, Norman TR, Eyre HA, Stahl SM, Phillips A, Carvalho AF, Berk M. Psilocybin in neuropsychiatry: a review of its pharmacology, safety, and efficacy. CNS Spectr. 2023 Aug;28(4):416-426. doi: 10.1017/S1092852922000888. Epub 2022 Jul 11. PMID 35811423
- [Background] Mertens LJ, Wall MB, Roseman L, Demetriou L, Nutt DJ, Carhart-Harris RL. Therapeutic mechanisms of psilocybin: Changes in amygdala and prefrontal functional connectivity during emotional processing after psilocybin for treatment-resistant depression. J Psychopharmacol. 2020 Feb;34(2):167-180. doi: 10.1177/0269881119895520. Epub 2020 Jan 16. PMID 31941394
- [Background] Goodwin GM, Aaronson ST, Alvarez O, Arden PC, Baker A, Bennett JC, Bird C, Blom RE, Brennan C, Brusch D, Burke L, Campbell-Coker K, Carhart-Harris R, Cattell J, Daniel A, DeBattista C, Dunlop BW, Eisen K, Feifel D, Forbes M, Haumann HM, Hellerstein DJ, Hoppe AI, Husain MI, Jelen LA, Kamphuis J, Kawasaki J, Kelly JR, Key RE, Kishon R, Knatz Peck S, Knight G, Koolen MHB, Lean M, Licht RW, Maples-Keller JL, Mars J, Marwood L, McElhiney MC, Miller TL, Mirow A, Mistry S, Mletzko-Crowe T, Modlin LN, Nielsen RE, Nielson EM, Offerhaus SR, O'Keane V, Palenicek T, Printz D, Rademaker MC, van Reemst A, Reinholdt F, Repantis D, Rucker J, Rudow S, Ruffell S, Rush AJ, Schoevers RA, Seynaeve M, Shao S, Soares JC, Somers M, Stansfield SC, Sterling D, Strockis A, Tsai J, Visser L, Wahba M, Williams S, Young AH, Ywema P, Zisook S, Malievskaia E. Single-Dose Psilocybin for a Treatment-Resistant Episode of Major Depression. N Engl J Med. 2022 Nov 3;387(18):1637-1648. doi: 10.1056/NEJMoa2206443. PMID 36322843